CLINICAL TRIAL: NCT01760486
Title: Using a State-wide Initiative to Disseminate Effective Behavioral Weight Loss Strategies
Brief Title: State-wide Health Approach to Increase Reach and Effectiveness: Study 3
Acronym: SHARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 211699-11; R18DK083248 (NIH)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2013-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shape Up Rhode Island (Active Comparator): Individuals who join Shape Up Rhode Island 2013, enter our research study, and lose 5% of their initial body weight during the first two months of Shape Up will be randomized to one of the three maintenance interventions. If randomized to this treatment arm, participants will receive periodic newsletters throughout the 12 month trial.
  Interventions: Behavioral: Shape Up Rhode Island
- Shape Up Rhode Island + Professional Coach + Incentives (Experimental): Individuals who join Shape Up Rhode Island 2013, enter our research study, and lose 5% of their initial body weight during the first two months of Shape Up will be randomized to one of the three maintenance interventions. If randomized to this treatment arm, participants will receive a professional weight loss coach and will be incentivized for submitting information to their coach and meeting weight goals.
  Interventions: Behavioral: Shape Up Rhode Island + Professional Coach + Incentives
- Shape Up Rhode Island + Peer Coach + Incentives (Experimental): Individuals who join Shape Up Rhode Island 2013, enter our research study, and lose 5% of their initial body weight during the first two months of Shape Up will be randomized to one of the three maintenance interventions. If randomized to this treatment arm, participants will receive a peer coach and will be incentivized for reporting to their coach and meeting weight goals.
  Interventions: Behavioral: Shape Up Rhode Island + Peer Coach + Incentives

INTERVENTIONS:
Behavioral: Shape Up Rhode Island
  Arms: Shape Up Rhode Island
Behavioral: Shape Up Rhode Island + Professional Coach + Incentives
  Arms: Shape Up Rhode Island + Professional Coach + Incentives
Behavioral: Shape Up Rhode Island + Peer Coach + Incentives
  Arms: Shape Up Rhode Island + Peer Coach + Incentives

SUMMARY:
The investigators have shown that adding an internet behavioral weight loss program to a statewide campaign improves weight loss outcomes. However, our follow-up data suggest that once the intervention is stopped, participants begin to experience weight regain. Thus, the purpose of this project is extend this line of work and pilot test health coaches and monetary incentives for weight loss maintenance. The investigators hypothesize that coaching and incentives will improve longer-term weight outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index >=25kg/m2
2. English speaking

Exclusion Criteria:

1. Health problems that make weight loss or unsupervised exercise unsafe
2. Current pregnancy or plan to become pregnant in the next 12 months
3. Planned relocation
4. Previous participation in Shape Up Rhode Island research studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
weight change from month 2 (i.e. immediately following the weight loss phase) to the 12 month follow-up assessment measured on a digital scale to the nearest 0.1 kilogram | 2 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States